CLINICAL TRIAL: NCT02268448
Title: Treatment of Chronic Itch in Atopic Dermatitis With Oral Clonidine and Oral Naltrexone: Nerve Function
Brief Title: Treatment of Chronic Itch in Atopic Dermatitis (Eczema): Nerve Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DERM-2006-15390
Record Dates: First submitted 2014-10-09; First posted 2014-10-20 (Estimated); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Cutaneous Nerves CNS Itch
Keywords: itch atopic dermatitis
MeSH Terms: interventions — Clonidine; Naltrexone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Clonidine (Experimental): Clonidine will be given orally as a starting dose of 0.1 mg daily. The drug will be administered orally by the subject at bedtime daily for four weeks.
  Interventions: Drug: Clonidine
- Naltrexone (Experimental): Naltrexone will be given to each subject at an oral dose of 50 mg daily. Subjects will self-administer the drug at bedtime.
  Interventions: Drug: Naltrexone

INTERVENTIONS:
Drug: Clonidine
  Arms: Clonidine
Drug: Naltrexone
  Arms: Naltrexone

SUMMARY:
The purpose of this study is to assess the safety and efficacy of oral clonidine in subjects with symptomatic atopic dermatitis and to assess the safety and efficacy of oral naltrexone in subjects with symptomatic atopic dermatitis.

DETAILED DESCRIPTION:
This study will serve as a pilot study to determine the efficacy and safety of two novel oral agents (clonidine, naltrexone) in the treatment of chronic, non-experimentally induced itch in atopic dermatitis. In this study, eight subjects with symptomatic atopic dermatitis will be recruited and treated with either oral clonidine (four subjects) or oral naltrexone (four subjects) . Disease burden will be evaluated before and after 4 weeks of treatment through reporting of subjective symptomatology via surveys/questionnaire, neurometer study, and clinical assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Age range 18-70 years old and ability to give informed consent and HIPAA authorization.
2. Female subjects of childbearing potential must have a negative pregnancy test, and must agree to practice two methods of effective birth control during the study period as clonidine is an FDA pregnancy category C drug (including abstinence, oral or implant contraceptives or condoms).
3. Diagnosis of AD via simplified UK Working Group Criteria and a baseline PSGA score of 2 or greater
4. Willingness to adhere to study protocol
5. Subjects taking hormone-containing medications must be on a stable dose for 6 months prior to study start to avoid any confounding influence on sensory and pain perception

Exclusion Criteria:

1. Use of topical or oral anti-inflammatory medications for 2 weeks prior to the study start.
2. Use of topical or oral anti-histamines for 2 weeks prior to the study start.
3. Use of topical or oral anti-pruritic agents for 2 weeks prior to the study start.
4. Use of oral neuromodulatory agents for 2 months prior to study start.
5. Current use of chronic pain medications (including opioids, antidepressants and anti-epileptic drugs).
6. Use of nicotine-containing products for the past 6 months prior to study start.
7. History of radiation or chemotherapy.
8. History of traumatic injury on prospective test sites.
9. Unstable thyroid function within the past 6 months prior to study start to exclude thyroid-related neuropathy (Duyff et al, 2000).
10. Known history of central or peripheral nervous system dysfunction.
11. History of acute hepatitis, chronic liver disease or end stage liver disease.
12. History of human immunodeficiency virus (HIV) or acquired immune deficiency syndrome.
13. History of neuropathy associated with chronic obstructive pulmonary disease, diabetes mellitus, documented exposure to organophosphates or heavy metals or polychlorinated biphenyls.
14. Known nutritional deficiency (vitamin B12, vitamin D, iron or zinc) within 3 months prior to the study start.
15. Use of illicit drugs within the past 6 months prior to study start.
16. History of daily use of power tools.
17. Lyme disease, porphyria, rheumatoid arthritis, Hansen's disease (leprosy) or use of antineoplastic chemotherapeutic agents.
18. Subject has any medical condition that, in the judgment of the Investigator, would jeopardize the subject's safety following exposure to the administered medications.
19. Adults lacking capacity to consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2022-09 (Actual); Study Completion 2022-09 (Actual)

PRIMARY OUTCOMES:
Reduction in Itch | 3 month
  Participants will take personal surveys regarding the reduction in itching after 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Maria Hordinsky, MD, Study Chair — University of Minnesota
Locations (1):
- University of Minnesota Department of Dermatology, Minneapolis, Minnesota, United States